CLINICAL TRIAL: NCT04575402
Title: Evaluating the Role of Wearable Technology and Patient-reported Outcomes to Monitor Physical Function Decline in Prostate Cancer Survivors
Brief Title: Digitally Captured Activity Data and PROs to Monitor Physical Function in Prostate Cancer Patients
Acronym: DigiPRO
Status: Active, not recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gillian Gresham, Assistant Professor, Cedars-Sinai Medical Center
Other Study IDs: IIT2020-15-GRESH-DIGIPRO
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Cancer survivorship; Wearable technology; Activity Monitors
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CSMC prostate cancer patients receiving ADT: Prostate cancer patients recruited from oncology clinic at Cedars-Sinai Medical Center.
  Interventions: Other: Wearable Activity Monitor
- Veterans with prostate cancer: Prostate cancer patients recruited from the Veteran Affairs Oncology Clinic (Durham, NC).
  Interventions: Other: Wearable Activity Monitor

INTERVENTIONS:
Other: Wearable Activity Monitor — Continuous monitoring of physical activity including step counts, sleep, heart rate, with consumer-based wearable activity monitor (Fitbit Charge HR4 or similar model)
  Other Names: Fitbit Charge HR; Wearable tracker; Wearable biosensor

SUMMARY:
Prospective observational research study to evaluate the role of wearable activity monitors to predict physical function decline among prostate cancer survivors receiving ADT.

DETAILED DESCRIPTION:
Physical function is a known predictor of QOL in advanced prostate cancer patients and key measure of treatment tolerability. While treatment with Androgen Deprivation Therapy (ADT) improves survival, it is associated with significant toxicities that lead to physical function (PF) decline. The average age of incident prostate cancer is 66 years, and in this older group of men, chronic comorbid conditions often co-occur with diagnosis, further adding to the risk for PF decline. With over 2.9 million prostate cancer survivors in the US, there is an increasing demand for adequate symptom monitoring and PF assessment throughout cancer care. However, there are currently no validated methods to systematically evaluate and predict PF decline. Thus, the overarching objective of this proposal is to determine whether the use of wearable technology to monitor objective daily activity combined with routine symptom reporting can predict PF decline. To accomplish this, we propose a mixed-methods approach that will provide quantitative information to help identify PC survivors at higher risk for PF decline as well as a qualitative aim gain a deeper understanding of the perceived relationships that PC survivors have with their physical activity levels and treatment symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients receiving ADT (+/- radiation) or planning to receive ADT. Start date of ADT must be planned for no more 7 days after baseline, or patients must have started ADT within 6 months prior to enrollment.
* 18 years or older
* Ambulatory (use of walking aids, such as cane and rollator, is acceptable)
* Access to a device that has the capability to sync to the Fitbit
* Have an understanding, ability, and willingness to fully comply with study procedures and restrictions
* English or Spanish speaking
* Informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

* Using a pacemaker, implantable cardiac defibrillator, neurostimulator, implantable hearing aids, cochlear implants, or other electronic medical equipment. However, removable hearing aids are permitted.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate cancer patients receiving ADT (+/- radiation) being seen for treatment at Cedars-Sinai Medical Center or the VA (Durham)
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-02-19 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical function decline within 3 months from baseline | 3 months
  Patient-reported physical function defined as 5-point change in standardized NIH PROMIS t-scores (mean 50, SD: 10), where higher scores represent higher physical function)
Absolute change in average step counts at 3 months from baseline | 3 months
  Change will be calculated based on difference in average weekly step count at baseline from the average weekly step count at end-of-study visit as measured using a Fitbit activity monitor where mean weekly Fitbit activity values will be calculated

SECONDARY OUTCOMES:
Mean change in Fitbit 24-hour activity | 3 months
  Change will be calculated based on difference in 24 hour activity as defined as periods of active minutes, sedentary time, and sleep at baseline and end-of-study
Key themes and concepts surrounding the relationships patients have with their treatment symptoms and how they affect their daily activity, as assessed in qualitative interviews. | 3 months
  This is a qualitative endpoint assessed in individual patient interviews at end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Gillian Gresham, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided